CLINICAL TRIAL: NCT00855595
Title: An Exploratory, Multicenter, Investigator-blinded, Active-controlled Study to Investigate the Efficacy of Topical Azelaic Acid (AzA)15% Gel Twice Daily or Metronidazole Topical Gel 1% Once Daily, Plus Anti-inflammatory Dose Doxycycline (40mg) Once Daily in Subjects With Moderate Papulopustular Rosacea
Brief Title: Efficacy of Topical Azelaic Acid 15% Gel Plus Anti-inflammatory Dose Doxycycline or Metronidazole Gel 1% Plus Anti-inflammatory Dose Doxycycline in Moderate Papulopustular Rosacea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14366; 1402604 (Other: Intendis GmbH); 256-0024 (Other: Intendis GmbH)
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Results first posted 2012-08-29 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2014-01

CONDITIONS: Papulopustular Rosacea
Keywords: Rosacea
MeSH Terms: conditions — Rosacea | interventions — azelaic acid; Metronidazole; Doxycycline

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azelaic acid (Finacea, BAY39-6251) plus Doxycycline (Oracea) (Experimental): Participants received topical azelaic acid gel 15% twice daily and doxycycline 40 mg once daily for 12 weeks
  Interventions: Drug: Azelaic acid (Finacea, BAY39-6251); Drug: Doxycycline (Oracea)
- Metronidazole (Metrogel) plus Doxycycline (Oracea) (Active Comparator): Participants received topical metronidazole 1% gel once daily and doxycycline 40 mg once daily for 12 weeks
  Interventions: Drug: Metronidazole (Metrogel); Drug: Doxycycline (Oracea)

INTERVENTIONS:
Drug: Azelaic acid (Finacea, BAY39-6251) — Participants received topical azelaic acid gel 15% twice daily for 12 weeks
  Arms: Azelaic acid (Finacea, BAY39-6251) plus Doxycycline (Oracea)
Drug: Metronidazole (Metrogel) — Participants received topical metronidazole 1% gel once daily for 12 weeks
  Arms: Metronidazole (Metrogel) plus Doxycycline (Oracea)
Drug: Doxycycline (Oracea) — Participants received systemic doxycycline 40 mg once daily for 12 week

SUMMARY:
Subjects with moderate papulopustular rosacea will be treated either with azelaic acid 15% gel topically plus an anti-inflammatory dose of doxycyline (40mg) daily or with metronidazole 1% gel topically once daily plus an anti-inflammatory dose of doxycycline (40mg) over at total of twelve weeks to determine the rapidity of improvement, and the length of time to reach 25%, 50% and 75% clearing compared to baseline.

DETAILED DESCRIPTION:
The change in inflammatory lesion count will be assessed at each post-baseline visit by an analysis of variance model (ANOVA) with factors treatment and center, but not including treatment-by-center interaction.

Investigator's Global Assessment (IGA) of papulopustular rosacea (static score): 0 - Clear (Virtually no rosacea ie, no papules and/or pustules; no or residual erythema; no or mild to moderate degree of telangiectasia may be present); 1 - Minimal (Rare papules and/or pustules; residual to mild erythema; mild to moderate degree of telangiectasia may be present); 2 - Mild (Few papules and/or pustules; mild erythema; mild to moderate degree of telangiectasia may be present); 3 - Mild to moderate (Distinct number of papules and/or pustules; mild to moderate erythema; mild to moderate degree of telangiectasia may be present); 4 - Moderate (Pronounced number of papules and/or pustules; moderate erythema; mild to moderate degree of telangiectasia may be present); 5 - Moderate to severe (Many papules and/or pustules, occasionally with large inflamed lesions; moderate erythema; moderate degree of telangiectasia may be present); 6 - Severe (Numerous papules and/or pustules, occasionally with confluent areas of inflamed lesions; moderate or severe erythema; moderate or severe degree of telangiectasia may be present).

ELIGIBILITY:
Inclusion Criteria:

- Moderate papulopustular rosacea (IGA>4) with a minimum of 10 and no more than 50 inflammatory lesions and persistent erythema with or without telangiectasia

Exclusion Criteria:

* Sensitivity to any of the treatments used
* Co-existing conditions that would unfavorably influence the course of the disease
* Pregnant or lactating women
* Severe rosacea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (17):
- United States (17):
  - Birmingham, Alabama
  - Denver, Colorado
  - West Palm Beach, Florida
  - Boston, Massachusetts
  - Warren, Michigan
  - Fridley, Minnesota
  - Henderson, Nevada
  - Albuquerque, New Mexico
  - Stony Brook, New York
  - Mason, Ohio
  - Portland, Oregon
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia

REFERENCES:
- [Result] Del Rosso JQ, Bruce S, Jarratt M, Menter A, Staedtler G. Efficacy of topical azelaic acid (AzA) gel 15% plus oral doxycycline 40 mg versus metronidazole gel 1% plus oral doxycycline 40 mg in mild-to-moderate papulopustular rosacea. J Drugs Dermatol. 2010 Jun;9(6):607-13. PMID 20645521

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) | Metronidazole (Metrogel) Plus Doxycycline (Oracea)
Started | 106 | 101
Completed | 100 | 94
Not Completed | 6 | 7
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 3 | 3
Not completed — Adverse Event | 1 | 1
Not completed — patient moved out of state | 1 | 0
Not completed — patient left country | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) | Metronidazole (Metrogel) Plus Doxycycline (Oracea) | Total
Number analyzed (Participants) | 106 | 101 | 207
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.4 (12.7) | 48.4 (11.5) | 49.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 69 | 136
  Male | 39 | 32 | 71
Investigator's Global Assessment (IGA) score at Baseline [Number; unit: Participants] — IGA categories: 0 - Clear; 1 - Minimal; 2 - Mild; 3 - Mild to moderate; 4 - Moderate; 5 - Moderate to severe; 6 - Severe (refer to Detailed Description field in Protocol section for more information).
  Participants
    IGA Score 4 - Moderate | 79 | 76 | 155
    IGA Score 5 - Moderate to Severe | 26 | 22 | 48
    IGA Score 6- Severe | 1 | 3 | 4
Number of lesions at Baseline [Mean (Standard Deviation); unit: Lesions] | 20.6 (11.01) | 21.9 (10.50) | 21.3 (10.76)
Previous duration of rosacea [Mean (Standard Deviation); unit: Months] | 130.8 (126.1) | 134.9 (107.2) | 132.8 (117.0)

OUTCOME MEASURES:

1. Primary Outcome: Nominal Change From Baseline in Inflammatory Lesion (IL) Count (Sum of Papules and Pustules) at Week 2 (LOCF: Last Observation Carried Forward)
Description: NOTE: Negative mean values represent an improvement (decrease of inflammatory lesions)
Time Frame: Baseline and Week 2
Population: Full analysis set (FAS)
Measure: Mean (Standard Deviation); unit: Inflammatory lesions
Arm/Group | Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) | Metronidazole (Metrogel) Plus Doxycycline (Oracea)
Number analyzed (Participants) | 106 | 101
Inflammatory lesions | -10.5 (9.14) | -9.4 (9.38)
Statistical Analysis 1: Comparison: Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) vs Metronidazole (Metrogel) Plus Doxycycline (Oracea); Test type: Superiority or Other; p = 0.0903, ANCOVA

2. Secondary Outcome: Number of Inflammatory Lesions at Weeks 2, 4, 6, 8 and 12 (LOCF)
Time Frame: Week 2, 4, 6, 8 and 12
Population: FAS
Measure: Mean (Standard Deviation); unit: Inflammatory lesions
Arm/Group | Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) | Metronidazole (Metrogel) Plus Doxycycline (Oracea)
Number analyzed (Participants) | 106 | 101
Inflammatory lesions
  Week 2 | 10.1 (8.70) | 12.5 (9.86)
  Week 4 | 7.4 (7.29) | 9.5 (8.09)
  Week 6 | 5.9 (6.28) | 7.8 (7.18)
  Week 8 | 5.1 (6.28) | 6.4 (7.02)
  Week 12 | 4.4 (6.51) | 5.7 (7.22)

3. Secondary Outcome: Nominal Change From Baseline in IL Count at Weeks 4, 6, 8 and 12 (LOCF)
Description: NOTE: Negative mean values represent an improvement (decrease of inflammatory lesions)
Time Frame: Baseline and Week 4, 6, 8 and 12
Population: FAS
Measure: Mean (Standard Deviation); unit: Inflammatory lesions
Arm/Group | Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) | Metronidazole (Metrogel) Plus Doxycycline (Oracea)
Number analyzed (Participants) | 106 | 101
Inflammatory lesions
  Week 4 | -13.2 (9.03) | -12.4 (9.23)
  Week 6 | -14.8 (9.20) | -14.1 (9.32)
  Week 8 | -15.5 (9.69) | -15.6 (9.82)
  Week 12 | -16.2 (9.88) | -16.2 (10.01)

4. Secondary Outcome: Percent Change From Baseline in IL Count at Weeks 2, 4, 6, 8 and 12 (LOCF)
Description: NOTE: Negative mean values represent an improvement (decrease of inflammatory lesions)
Time Frame: Baseline and Week 2, 4, 6, 8 and 12
Population: FAS
Measure: Mean (Standard Deviation); unit: Percent of inflammatory lesions
Arm/Group | Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) | Metronidazole (Metrogel) Plus Doxycycline (Oracea)
Number analyzed (Participants) | 106 | 101
Percent of inflammatory lesions
  Week 2 | -50.7 (29.39) | -43.0 (35.68)
  Week 4 | -64.9 (28.93) | -56.9 (31.50)
  Week 6 | -72.4 (24.67) | -64.5 (29.00)
  Week 8 | -76.4 (23.47) | -71.6 (26.94)
  Week 12 | -80.2 (24.25) | -75.1 (27.25)

5. Secondary Outcome: Percentage of Participants With at Least a 25%, 50%, or 75% Improvement in Facial IL Counts From Baseline to Weeks 2, 4, 6, 8 and 12 (LOCF)
Time Frame: Baseline and Weeks 2, 4, 6, 8 and 12
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) | Metronidazole (Metrogel) Plus Doxycycline (Oracea)
Number analyzed (Participants) | 106 | 101
Percentage of participants
  Week 2, ≥25% improvement | 84.9 | 77.2
  Week 2, ≥50% improvement | 61.3 | 47.5
  Week 2, ≥75% improvement | 20.8 | 17.8
  Week 4, ≥25% improvement | 90.6 | 81.2
  Week 4, ≥50% improvement | 75.5 | 64.4
  Week 4, ≥75% improvement | 44.3 | 40.6
  Week 6, ≥25% improvement | 95.3 | 91.1
  Week 6, ≥50% improvement | 84.9 | 78.2
  Week 6, ≥75% improvement | 54.7 | 43.6
  Week 8, ≥25% improvement | 95.3 | 90.1
  Week 8, ≥50% improvement | 88.7 | 87.1
  Week 8, ≥75% improvement | 67.0 | 55.4
  Week 12, ≥25% improvement | 96.2 | 91.1
  Week 12, ≥50% improvement | 89.6 | 85.1
  Week 12, ≥75% improvement | 68.9 | 65.3

6. Secondary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Based Therapeutic Success at Weeks 2, 4, 6, 8 and 12 (LOCF)
Description: IGA categories: 0 - Clear; 1 - Minimal; 2 - Mild; 3 - Mild to moderate; 4 - Moderate; 5 - Moderate to severe; 6 - Severe (refer to Detailed Description field in Protocol section for more information) / Therapeutic success is defined as an IGA score of clear or minimal (0 or 1).
Time Frame: Weeks 2, 4, 6, 8 and 12
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) | Metronidazole (Metrogel) Plus Doxycycline (Oracea)
Number analyzed (Participants) | 106 | 101
Percentage of participants
  Week 2 | 13.2 | 7.9
  Week 4 | 32.1 | 26.7
  Week 6 | 45.3 | 27.7
  Week 8 | 50.9 | 39.6
  Week 12 | 62.3 | 52.5

7. Secondary Outcome: Percentage of Participants With IGA Based Patient Response at Weeks 2, 4, 6, 8 and 12 (LOCF)
Description: IGA categories: 0 - Clear; 1 - Minimal; 2 - Mild; 3 - Mild to moderate; 4 - Moderate; 5 - Moderate to severe; 6 - Severe (refer to Detailed Description field in Protocol section for more information) / Patient response is defined as an IGA score of clear, minimal, or mild (0, 1, or 2)
Time Frame: Weeks 2, 4, 6, 8 and 12
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) | Metronidazole (Metrogel) Plus Doxycycline (Oracea)
Number analyzed (Participants) | 106 | 101
Percentage of participants
  Week 2 | 32.1 | 27.7
  Week 4 | 55.7 | 44.6
  Week 6 | 60.4 | 53.5
  Week 8 | 72.6 | 59.4
  Week 12 | 78.3 | 72.3

8. Secondary Outcome: Percentage of Participants With Respective Disease Severity Measured by IGA Scores at Week 2
Description: IGA categories: 0 - Clear; 1 - Minimal; 2 - Mild; 3 - Mild to moderate; 4 - Moderate; 5 - Moderate to severe; 6 - Severe (refer to Detailed Description field in Protocol section for more information).
Time Frame: At Week 2
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) | Metronidazole (Metrogel) Plus Doxycycline (Oracea)
Number analyzed (Participants) | 106 | 101
Percentage of participants
  0 - Clear | 0.9 | 1.0
  1 - Minimal | 12.3 | 6.9
  2 - Mild | 18.9 | 19.8
  3 - Mild to moderate | 33.0 | 31.7
  4 - Moderate | 25.5 | 27.7
  5 - Moderate to severe | 9.4 | 10.9
  6 - Severe | 0 | 2.0

9. Secondary Outcome: Percentage of Participants With Respective Disease Severity Measured by IGA Scores at Week 4
Description: as for outcome 8
Time Frame: At Week 4
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) | Metronidazole (Metrogel) Plus Doxycycline (Oracea)
Number analyzed (Participants) | 106 | 101
Percentage of participants
  0 - Clear | 7.5 | 6.9
  1 - Minimal | 24.5 | 19.8
  2 - Mild | 23.6 | 17.8
  3 - Mild to moderate | 24.5 | 23.8
  4 - Moderate | 15.1 | 20.8
  5 - Moderate to severe | 4.7 | 9.9
  6 - Severe | 0 | 1.0

10. Secondary Outcome: Percentage of Participants With Respective Disease Severity Measured by IGA Scores at Week 6
Description: as for outcome 8
Time Frame: At Week 6
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) | Metronidazole (Metrogel) Plus Doxycycline (Oracea)
Number analyzed (Participants) | 106 | 101
Percentage of participants
  0 - Clear | 18.9 | 9.9
  1 - Minimal | 26.4 | 17.8
  2 - Mild | 15.1 | 25.7
  3 - Mild to moderate | 24.5 | 19.8
  4 - Moderate | 11.3 | 19.8
  5 - Moderate to severe | 3.8 | 6.9
  6 - Severe | 0 | 0

11. Secondary Outcome: Percentage of Participants With Respective Disease Severity Measured by IGA Scores at Week 8
Description: as for outcome 8
Time Frame: At Week 8
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) | Metronidazole (Metrogel) Plus Doxycycline (Oracea)
Number analyzed (Participants) | 106 | 101
Percentage of participants
  0 - Clear | 18.9 | 13.9
  1 - Minimal | 32.1 | 25.7
  2 - Mild | 21.7 | 19.8
  3 - Mild to moderate | 14.2 | 23.8
  4 - Moderate | 10.4 | 12.9
  5 - Moderate to severe | 2.8 | 4.0
  6 - Severe | 0 | 0

12. Secondary Outcome: Percentage of Participants With Respective Disease Severity Measured by IGA Scores at Week 12
Description: as for outcome 8
Time Frame: At Week 12
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) | Metronidazole (Metrogel) Plus Doxycycline (Oracea)
Number analyzed (Participants) | 106 | 101
Percentage of participants
  0 - Clear | 30.2 | 22.8
  1 - Minimal | 32.1 | 29.7
  2 - Mild | 16.0 | 19.8
  3 - Mild to moderate | 12.3 | 13.9
  4 - Moderate | 6.6 | 10.9
  5 - Moderate to severe | 1.9 | 3.0
  6 - Severe | 0.9 | 0

13. Secondary Outcome: Investigator Rating of Overall Improvement at End of Study (Week 12)
Time Frame: Week 12
Population: Participants in the FAS who took part in this evaluation.
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) | Metronidazole (Metrogel) Plus Doxycycline (Oracea)
Number analyzed (Participants) | 103 | 97
Percentage of participants
  Excellent Improvement | 46.6 | 42.3
  Marked Improvement | 35.9 | 34.0
  Moderate Improvement | 12.6 | 17.5
  No change | 4.9 | 6.2
  Deterioration | 0 | 0

14. Secondary Outcome: Patient Rating of Overall Improvement at End of Study (Week 12)
Time Frame: Week 12
Population: Participants in the FAS who took part in this evaluation.
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) | Metronidazole (Metrogel) Plus Doxycycline (Oracea)
Number analyzed (Participants) | 102 | 96
Percentage of participants
  Excellent Improvement | 51.0 | 49.0
  Good Improvement | 39.2 | 33.3
  Fair Improvement | 7.8 | 15.6
  No Improvement | 2.0 | 1.0
  Worse | 0 | 1.0

15. Secondary Outcome: Patient Opinion of Cosmetic Acceptability at End of Study (Week 12)
Time Frame: Week 12
Population: Participants in the FAS who took part in this evaluation.
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) | Metronidazole (Metrogel) Plus Doxycycline (Oracea)
Number analyzed (Participants) | 102 | 96
Percentage of participants
  Very Good | 52.0 | 56.3
  Good | 34.3 | 26.0
  Satisfactory | 4.9 | 8.3
  Poor | 0 | 1.0
  No Opinion | 8.8 | 8.3

16. Other Pre Specified Outcome: Patient Opinion of Local Tolerability
Time Frame: Week 12
Population: Participants in the FAS who took part in this evaluation.
Measure: Number; unit: Percentage of Participants
Arm/Group | Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) | Metronidazole (Metrogel) Plus Doxycycline (Oracea)
Number analyzed (Participants) | 102 | 96
Percentage of Participants
  Excellent | 53.9 | 72.9
  Good | 34.3 | 15.6
  Acceptable despite minor irritation | 7.8 | 11.5
  Less acceptable due to continuous irritation | 2.9 | 0
  No opinion | 1.0 | 0

ADVERSE EVENTS:
Groups:
- Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea): Participants received topical azelaic acid gel 15% twice daily and systemic doxycycline 40 mg once daily for 12 weeks
- Metronidazole (Metrogel) Plus Doxycycline (Oracea): Participants received topical metronidazole 1% gel once daily and systemic doxycycline 40 mg once daily for 12 weeks
Arm/Group | Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) | Metronidazole (Metrogel) Plus Doxycycline (Oracea)
Serious Adverse Events (participants affected / at risk) | 0/106 | 1/101
Other Adverse Events (participants affected / at risk) | 29/106 | 33/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) (N=106) | Metronidazole (Metrogel) Plus Doxycycline (Oracea) (N=101)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azelaic Acid (Finacea, BAY39-6251) Plus Doxycycline (Oracea) (N=106) | Metronidazole (Metrogel) Plus Doxycycline (Oracea) (N=101)
Ear congestion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (3)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Application site oedema (General disorders) | 0 (0) | 1 (1)
Application site pruritus (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Application site urticaria (General disorders) | 0 (0) | 1 (1)
Application site exfoliation (General disorders) | 0 (0) | 3 (7)
Application site burn (General disorders) | 1 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 4 (4) | 4 (4)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0)
Food poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 5 (8)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Elective surgery (Surgical and medical procedures) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A) Investigator shall provide Sponsor with intended publication 60 days upfront publication date, Sponsor has 30 d to comment, recommended changes shall not be unreasonably refused B) Sponsor has the right to ask Investigator to delay publication for a maximum of 90 days C) Investigative data will be pooled and published by Sponsor - no other publication without the consent of all parties prior to publication of the pooled data, or within 12 months after LPLV, whatever comes first